CLINICAL TRIAL: NCT02461459
Title: Autism Spectrum Disorder (ASD) and Intellectual Disability (ID) Determinants in Tuberous Sclerosis Complex (TSC)
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Tuberous Sclerosis Alliance (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Office of Rare Diseases (ORD) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mustafa Sahin, Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: IRB-P00013585; 1U54NS092090 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-06-03 (Estimated); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Tuberous Sclerosis; Autism Disorder; Intellectual Disability
Keywords: Tuberous Sclerosis Complex; TSC; Autism; ASD; Intellectual Disability; ID; MRI; EEG
MeSH Terms: conditions — Tuberous Sclerosis; Autistic Disorder; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw for future correlative studies in the TSC Biorepository of the Developmental Synaptopathies Consortium.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tuberous Sclerosis Complex: Tuberous Sclerosis Complex

SUMMARY:
The purpose of this study is to characterize the developmental phenotype of ASD and ID and to identify biomarkers using advanced MRI methodology and electrophysiological biomarkers of synaptic function and connectivity predictive of ASD and ID presence and severity in patients with TSC. In addition, this study will be establishing infrastructure for the collection and storage of human bio-specimens, including genetic material, from TSC patients and their family members with ASD.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is a multi-system disease that usually exhibits a high variability in clinical findings both among and within families. About 50% of individuals with TSC develop intellectual disability (ID) and/or autism spectrum disorder (ASD). The purpose of this research study is to learn more information about ASD/ID in individuals with TSC through neurobehavioral assessments, electroencephalogram (EEG) data, and magnetic resonance imaging so that ultimately effective treatments and interventions for ASD/ID can be realized.

Individuals with TSC will be asked to participate in this study if they are 18 months or older at the time of enrollment and have been diagnosed with suspected or confirmed autism spectrum disorder and/or intellectual disability, as well as healthy controls. Both males and females will be asked to participate. Additionally, to be eligible for study participation, individuals' primary communicative language must be English. The participant and at least one biological parent will be asked to provide biological specimens including DNA and RNA for inclusion in the TSC RDCRN Biorepository.

The study involves 3 on site visits over the course of two years. Study visits will vary in length from about 4 hours to 6 hours. Study visits involve a physical exam, medical history questions, and neuropsychological assessments. A subset of participants between the ages of 2 and 11 years old will take part in the EEG portion of the study. At one point during the study, a blood draw will be done for future research studies. Individuals who have a clinically indicated MRI will have an option to provide routine clinical scans for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Meets genetic or clinical diagnostic criteria for TSC (Tuberous Sclerosis), the latter based on current recommendations for diagnostic evaluation, such as physical exam, neuroimaging, and echocardiogram.
* Age criteria: over 18 months of age at time of enrollment.
* Is diagnosed or suspected to have ASD and/or ID.
* Primary communicative language is English

Exclusion Criteria:

* Has taken an investigational drug as part of another research study, within 30 days prior to study enrollment.
* For subjects involved in imaging biomarker assessment: contraindications to 3T MRI scanning, such as metal implants/non-compatible medical devices or medical conditions, including vagus nerve stimulator.
* For subjects involved in EEG/ERP biomarker assessment: contraindications to EEG/ERP, such as uncooperative or destructive behaviors preventing lead placement or capture by ERP/VEP equipment. Under age 2 or above age 11 at the time of enrollment.
* Unwilling or unable to comply with study procedures and assessments.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 195 participants over the age of 18 months old with TSC and suspected or diagnosed ASD, ID, or combined ASD/ID will be enrolled into the study. Diagnosis of TSC will be based on established clinical or genetic criteria. Subjects will be enrolled from current and new TSC patients at each of the 6 centers.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2015-05; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in ADOS-2 scores at end of study | 24 months
  Using standardized composite score for ADOS-2 performed yearly to determine ASD
Change in SBIS-5 scores or Mullen Scales of Early Learning (MSEL) at end of study | 24 months
  Using standardized IQ score from the Stanford-Binet Intelligence Scales Fifth Edition (SBIS-5) or Mullen Scales of Early Learning (MSEL) performed yearly to determine ID
Change in Fractional anisotropy (FA) at 12 months | 12 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be fractional anisotropy (FA) determined by MRI diffusion tensor imaging (DTI) with tractography at 12 months radial diffusivity (RD), axial diffusivity (AD), and mean diffusivity (MD) of cerebellar fascicles corresponding to the neuroanatomically-defined excitatory and inhibitory projections cerebellar Purkinje neurons,
Change in fractional anisotropy (FA) at 24 months | 24 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be fractional anisotropy (FA) determined by MRI diffusion tensor imaging (DTI) with tractography at 24 months
Change in radial diffusivity (RD) at 12 months | 12 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be radial diffusivity (RD) determined by MRI diffusion tensor imaging (DTI) with tractography at 12 months
Change in radial diffusivity (RD) at 24 months | 24 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be radial diffusivity (RD) determined by MRI diffusion tensor imaging (DTI) with tractography at 24 months
Change in mean diffusivity (MD) of cerebellar fascicles at 12 months | 12 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be mean diffusivity (MD) of cerebellar fascicles determined by MRI diffusion tensor imaging (DTI) with tractography at 12 months
Change in mean diffusivity (MD) of cerebellar fascicles at 24 months | 24 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be mean diffusivity (MD) of cerebellar fascicles determined by MRI diffusion tensor imaging (DTI) with tractography at 24 months
Change in axial diffusivity (AD) at 12 months | 12 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be axial diffusivity (AD) determined by MRI diffusion tensor imaging (DTI) with tractography at 12 months
Change in axial diffusivity (AD) at 24 months | 24 months
  To determine cerebellum white matter structural integrity, the primary outcome measures will be axial diffusivity (AD) determined by MRI diffusion tensor imaging (DTI) with tractography at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Krueger, MD, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas at Houston, Houston, Texas